CLINICAL TRIAL: NCT00004409
Title: Phase II Randomized Study of Collagenase in Patients With Residual Type Dupuytren's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13297; SUNY-SB-FDR001373; DUPY-101; DUPY-202; SUNY-SB-431-1007A; SUNY-SB-431-8804B; SUNY-SB-431-X2020
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-05

CONDITIONS: Dupuytren's Contracture
Keywords: Dupuytren's disease; arthritis & connective tissue diseases; rare disease
MeSH Terms: conditions — Dupuytren Contracture; Arthritis; Connective Tissue Diseases; Rare Diseases | interventions — Collagenases

INTERVENTIONS:
Drug: collagenase

SUMMARY:
OBJECTIVES:

Evaluate the safety and efficacy of collagenase in improving flexion deformity, range of motion, and grip strength in patients with residual Dupuytren's disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, investigator-blinded, placebo-controlled study.

Patients receive a single dose of either collagenase or placebo into the target finger on day 0. Patients who do not respond at the 1 month follow up visit may receive an injection of open label collagenase, if IgE antibody levels are no greater than 15 ng/mL.

Following treatment, patients use a nighttime extension splint for 4 months and perform finger flexion/extension exercises. Patients are followed at 1, 7, and 14 days, and at 1, 2, 3, 6, 9, and 12 months, for each joint treated.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Diagnosis of residual Dupuytren's disease with fixed flexion deformity of the fingers of at least 20-30 degrees caused by a palpable cord Positive table top test (inability to simultaneously place affected finger and palm flat against a table top) --Prior/Concurrent Therapy-- Surgery: At least 30 days since surgery for Dupuytren's disease Other: At least 30 days since prior investigational drug --Patient Characteristics-- Hematopoietic: No history of hematologic disease Hepatic: No history of hepatic disease Renal: No history of renal disease Cardiovascular: No congestive heart failure within 6 months No angina within 6 months No myocardial infarction within 6 months Pulmonary: No history of respiratory disease Other: HIV negative Not immunocompromised No history of significant illness, e.g., endocrine or neurologic disease No history of illicit drug abuse or alcoholism within 1 year No psychosis At least 2 weeks since infectious illness No chronic or debilitating disease No IgE antibodies to collagenase greater than 15 ng/mL No known allergy to collagenase or any of the inactive ingredients in the injection Not pregnant or nursing Fertile patients must use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 1995-08; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C. Hurst, Study Chair — State University of New York
Locations (2):
- United States (2):
  - Stanford University Hospital, Palo Alto, California
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York